CLINICAL TRIAL: NCT01213043
Title: A Randomized Double-blind Crossover Study to Assess the Safety and Pharmacokinetics of Two Different Doses of Weekly Intravenous Administration of Alpha1-Proteinase Inhibitor (Human) Prolastin®-C in Subjects With Alpha1-Antitrypsin Deficiency
Brief Title: Safety and Pharmacokinetics of Alpha-1 Proteinase Inhibitor in Subjects With Alpha1-Antitrypsin Deficiency
Acronym: SPARK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grifols Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: T6004-201/Version 2
Record Dates: First submitted 2010-09-29; First posted 2010-10-01 (Estimated); Results first posted 2013-05-20 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2013-04

CONDITIONS: Emphysema; Alpha 1-antitrypsin Deficiency (AATD)
Keywords: emphysema; alpha 1-antitrypsin; alpha 1-antitrypsin deficiency (AATD); alpha 1-proteinase inhibitor (Alpha-1 PI)
MeSH Terms: conditions — Emphysema; alpha 1-Antitrypsin Deficiency | interventions — alpha 1-Antitrypsin; Mp alpha1 receptor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prolastin-C, 60 mg/kg (Active Comparator): 60 mg/kg weekly infusion of Prolastin-C for 8 weeks. Subjects were infused with 60 mg/kg Prolastin-C by means of one of two possible treatment sequences: 1) 60 mg/kg weekly infusion of Prolastin-C for 8 weeks followed by 120 mg/kg Prolastin-C for 8 weeks, or 2) 120 mg/kg Prolastin-C for 8 weeks followed by 60 mg/kg weekly infusion of Prolastin-C for 8 weeks (total of 16 weeks).
  Interventions: Biological: Prolastin-C, 60 mg/kg
- Prolastin-C, 120 mg/kg (Experimental): 120 mg/kg weekly infusion of Prolastin-C for 8 weeks. Subjects were infused with 120 mg/kg Prolastin-C by means of one of two possible treatment sequences: 1) 60 mg/kg weekly infusion of Prolastin-C for 8 weeks followed by 120 mg/kg Prolastin-C for 8 weeks, or 2) 120 mg/kg Prolastin-C for 8 weeks followed by 60 mg/kg weekly infusion of Prolastin-C for 8 weeks (total of 16 weeks).
  Interventions: Biological: Prolastin-C, 120 mg/kg

INTERVENTIONS:
Biological: Prolastin-C, 60 mg/kg — 60 mg/kg weekly infusion of Prolastin-C for 8 weeks
  Other Names: Alpha1-Proteinase Inhibitor; Alpha1-Proteinase Inhibitor (Human), Modified Process; Alpha-1 MP
  Arms: Prolastin-C, 60 mg/kg
Biological: Prolastin-C, 120 mg/kg — 120 mg/kg weekly infusion of Prolastin-C for 8 weeks
  Other Names: Alpha1-Proteinase Inhibitor; Alpha1-Proteinase Inhibitor (Human), Modified Process; Alpha-1 MP
  Arms: Prolastin-C, 120 mg/kg

SUMMARY:
This is a study to assess the safety and pharmacokinetics of weekly infusions of 120 mg/kg of Prolastin-C (alpha1-proteinase inhibitor [alpha1-PI] [Human]), compared to weekly infusions of 60 mg/kg of Prolastin-C in patients with alpha 1-antitrypsin deficiency (AATD).

DETAILED DESCRIPTION:
The question of whether higher doses of alpha1-PI (>60 mg/kg) are able to provide better protection to patients with alpha 1-antitrypsin deficiency is currently unknown. As a first step to address this question, the present study has been undertaken. This is a multi-center, randomized, double-blind, crossover study to assess the safety and pharmacokinetics of weekly infusions of 120 mg/kg of Prolastin-C, compared to weekly infusions of 60 mg/kg of Prolastin-C in patients with alpha 1-antitrypsin deficiency. This study is a crossover design with 2 treatment sequences:

Treatment Sequence 1: 60 mg/kg weekly infusion of Prolastin-C for 8 weeks followed by 120 mg/kg weekly infusion of Prolastin-C for 8 weeks (starting at Week 1) (total of 16 treatment weeks)

Treatment Sequence 2: 120 mg/kg weekly infusion of Prolastin-C for 8 weeks followed by 60 mg/kg weekly infusion of Prolastin-C for 8 weeks (starting at Week 11) (total of 16 treatment weeks)

Approximately 15 subjects are planned to be entered into each treatment sequence.

At Weeks 8 to 11 and Weeks 18 to 21, a total of 15 serial blood samples for each subject will be drawn for pharmacokinetic analysis. The expected duration of the study subject's participation will be approximately 25 weeks (which includes a 3-Week Screening Phase, 2-Week Washout Period [between different alpha-1 PI treatment doses], and a 4-Week Follow-up Period). The following safety parameters will be assessed: adverse events, pulmonary exacerbations, vital signs, pulmonary function tests, and clinical laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

* Be between 18 and 70 years of age
* Have a documented diagnosis of congenital AATD
* Have a post-bronchodilator Forced Expired Volume in 1 second (FEV1) of ≥30% and <80% and FEV1/forced vital capacity (FVC) <70%
* If receiving alpha-1 PI augmentation therapy, be willing to discontinue the treatment for the duration of the study

Exclusion Criteria:

* Had a moderate or severe pulmonary exacerbation during the 4 weeks before the study
* History of lung or liver transplant
* Any lung surgery during the past 2 years
* Confirmed liver cirrhosis
* Elevated liver enzymes
* Severe concurrent disease
* Females who are pregnant or breast-feeding or unwilling to practice effective contraception during the study
* Infection with hepatitis A, B, or C, human immunodeficiency or parvovirus B19
* Smoking during the past 6 months
* Use of systemic steroids within 4 weeks of the study
* Use of antibiotics for an exacerbation within 4 weeks of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Brantly, MD, Principal Investigator — University of Florida; Michael Campos, MD, Principal Investigator — University of Miami; Friedrich Kueppers, MD, Principal Investigator — Temple University Hospital/Temple Lung Center; James Stocks, MD, Principal Investigator — The University of Texas Health Science Center at Tyler; Charlie Strange, MD, Principal Investigator — Medical University of South Carolina, Division of Pulmonary and Critical Care Medicine
Locations (5):
- United States (5):
  - University of Florida College of Medicine, Gainesville, Florida
  - University of Miami, Miami, Florida
  - Temple University Hosptial/Temple Lung Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Division of Pulmonary and Critical Care Medicine, Charleston, South Carolina
  - The University of Texas Health Science Center at Tyler, Tyler, Texas

REFERENCES:
- [Background] Willis T, Wee K, Mohn G. A high-purity Alpha-1 proteinase inhibitor from human plasma, TAL6004. Proceeding of the 19th European Respiratory Society Annual Congress; 2009 Sep 12-16; Vienna, Austria. Abstracts;34:S53.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects entered a Screening Phase (up to 21 days in duration) to determine subject eligibility and for wash-out of prior alpha1-PI augmentation therapy, if applicable, prior to randomization to one of two treatment sequences.
Groups:
- 60 mg/kg - 120 mg/kg Prolastin-C Treatment Sequence: Weekly infusions of 60 mg/kg Prolastin-C for 8 weeks followed by a 2-week off-treatment washout period followed by weekly infusions of 120 mg/kg Prolastin-C for 8 weeks (total of 16 treatment weeks)
- 120 mg/kg - 60 mg/kg Prolastin-C Treatment Sequence: Weekly infusions of 120 mg/kg Prolastin-C for 8 weeks followed by a 2-week off-treatment washout period followed by weekly infusions of 60 mg/kg Prolastin-C for 8 weeks (total of 16 treatment weeks)
Period: Treatment Period 1
Arm/Group | 60 mg/kg - 120 mg/kg Prolastin-C Treatment Sequence | 120 mg/kg - 60 mg/kg Prolastin-C Treatment Sequence
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: Washout Period
Arm/Group | 60 mg/kg - 120 mg/kg Prolastin-C Treatment Sequence | 120 mg/kg - 60 mg/kg Prolastin-C Treatment Sequence
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: Treatment Period 2
Arm/Group | 60 mg/kg - 120 mg/kg Prolastin-C Treatment Sequence | 120 mg/kg - 60 mg/kg Prolastin-C Treatment Sequence
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: Follow-up
Arm/Group | 60 mg/kg - 120 mg/kg Prolastin-C Treatment Sequence | 120 mg/kg - 60 mg/kg Prolastin-C Treatment Sequence
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Demographic and other baseline characteristics were analyzed on the intent-to-treat population, which included all subjects who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | 60 mg/kg - 120 mg/kg Prolastin-C Treatment Sequence | 120 mg/kg - 60 mg/kg Prolastin-C Treatment Sequence | Total
Number analyzed (Participants) | 15 | 15 | 30
Age Continuous [Mean (Standard Deviation); unit: years] | 59.7 (6.89) | 57.4 (6.34) | 58.6 (6.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 7 | 7 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 15 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Subjects With Treatment-Emergent Adverse Events (TEAEs)
Description: Number of subjects experiencing at least one TEAE. TEAEs were defined as any adverse event (AE) during the study that began on or after the date of first dose of investigational product (i.e., Prolastin-C).
Time Frame: 22 weeks
Population: All safety analyses were performed on the safety population, which comprised of all subjects who were randomized and received at least one dose of investigational product (Prolastin-C).
Measure: Number; unit: participants
Arm/Group | 60 mg/kg Prolastin-C | 120 mg/kg Prolastin-C
Number analyzed (Participants) | 30 | 30
participants | 23 | 18

2. Secondary Outcome: AUC0-7days
Description: Area Under the Alpha-1 PI Concentration-Time Curve from Day 0 to Day 7
Time Frame: Week 8 and Week 18 at the following timepoints: 0 (pre-infusion), completion of first infusion bag, completion of 2nd infusion bag, and 15 min, 30 min, and 1, 2, 4, 8, 24, 48, 120, and 168 hours post-dose
Population: Pharmacokinetic (PK) Population, which consisted of all subjects who received investigational product (Prolastin-C) and had sufficient and valid serum concentration data to facilitate calculation of PK parameters.
Measure: Mean (Standard Deviation); unit: h*mg/mL
Arm/Group | 60 mg/kg Prolastin-C | 120 mg/kg Prolastin-C
Number analyzed (Participants) | 29 | 30
h*mg/mL | 203.6 (20.48) | 344.8 (46.53)
Statistical Analysis 1: Comparison: 60 mg/kg Prolastin-C vs 120 mg/kg Prolastin-C; Dose proportionality was analysed using an ANOVA model for the natural log-transformed AUC0-7days with treatment, period, and sequence as fixed effects and subject within sequence as a random effect. The treatment dose of 60 mg/kg was the reference treatment and 120 mg/kg was the test treatment. PK parameters in individual subjects for each treatment dose were dose normalized to 60mg/kg based on the actual dose administered at Week 8 or Week 18 (i.e., (AUC0-7days/Actual Dose in mg/kg)*60mg/kg); Test type: Non-Inferiority or Equivalence — Equivalence margin was: [0.80, 1.25]; p < 0.0001, ANOVA; Geometric Least Square Means Ratio = 0.85, 90% CI 2-sided [0.83 to 0.88]

3. Primary Outcome: Subjects With Drug-Related TEAE(s)
Description: Number of subjects with at least one TEAE that was determined by the Investigator to be either "possibly related" or "related" to the investigational product (i.e., Prolastin-C).
Time Frame: 22 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | 60 mg/kg Prolastin-C | 120 mg/kg Prolastin-C
Number analyzed (Participants) | 30 | 30
participants | 3 | 1

4. Primary Outcome: Subjects With Treatment-Emergent Serious Adverse Events (SAEs)
Description: Number of subjects who experienced at least one treatment-emergent SAE.
Time Frame: 22 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | 60 mg/kg Prolastin-C | 120 mg/kg Prolastin-C
Number analyzed (Participants) | 30 | 30
participants | 0 | 0

5. Primary Outcome: Subjects Withdrawn Due to an AE(s)
Description: Number of subjects who were withdrawn from the study due to at least one AE.
Time Frame: 22 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | 60 mg/kg Prolastin-C | 120 mg/kg Prolastin-C
Number analyzed (Participants) | 30 | 30
participants | 0 | 0

6. Primary Outcome: Subjects With Treatment-Emergent Pulmonary Exacerbation(s)
Description: Number of subjects with at least one treatment-emergent pulmonary exacerbation
Time Frame: 22 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | 60 mg/kg Prolastin-C | 120 mg/kg Prolastin-C
Number analyzed (Participants) | 30 | 30
participants | 7 | 5

7. Primary Outcome: Subjects With Severe TEAE(s) or Pulmonary Exacerbation(s)
Description: Number of subjects who experienced at least one severe TEAE or pulmonary exacerbation.
Time Frame: 22 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | 60 mg/kg Prolastin-C | 120 mg/kg Prolastin-C
Number analyzed (Participants) | 30 | 30
participants | 0 | 0

8. Secondary Outcome: Mean Trough
Description: The average trough concentration at steady-state, calculated as the mean value using the four Trough measurements obtained at Weeks 6, 7, 8 and at 7 days (168 hours) post infusion at Week 8 for the first treatment period or prior to the start of the infusions at Weeks 16, 17, 18, and at 7 days (168 hours) post infusion at Week 18 for the second treatment period.
Time Frame: Single measurment immediately prior to infusion at Weeks 6, 7, 8, 9 and Weeks 16, 17, 18, 19
Population: PK Population, which consisted of all subjects who received investigational product (Prolastin-C) and had sufficient and valid serum concentration data to facilitate calculation of PK parameters.
Measure: Mean (Standard Deviation); unit: μM
Arm/Group | 60 mg/kg Prolastin-C | 120 mg/kg Prolastin-C
Number analyzed (Participants) | 30 | 30
μM | 17.3 (2.36) | 27.7 (3.75)

9. Primary Outcome: Number of TEAEs
Description: Total number of TEAEs reported.
Time Frame: 22 Weeks
Population: as for outcome 1
Measure: Number; unit: Events
Arm/Group | 60 mg/kg Prolastin-C | 120 mg/kg Prolastin-C
Number analyzed (Participants) | 30 | 30
Events | 69 | 43

10. Primary Outcome: Number of Drug-related TEAEs
Description: Total number of drug-related TEAEs reported
Time Frame: 22 Weeks
Population: as for outcome 1
Measure: Number; unit: Events
Arm/Group | 60 mg/kg Prolastin-C | 120 mg/kg Prolastin-C
Number analyzed (Participants) | 30 | 30
Events | 5 | 1

11. Primary Outcome: Number of Treatment-Emergent Pulmonary Exacerbations
Description: Total number of treatment-emergent pulmonary exacerbations.
Time Frame: 22 Weeks
Population: as for outcome 1
Measure: Number; unit: Events
Arm/Group | 60 mg/kg Prolastin-C | 120 mg/kg Prolastin-C
Number analyzed (Participants) | 30 | 30
Events | 9 | 6

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the time of informed consent through the end of study visit; thus, AEs were assessed for up to 25 weeks.
Description: Assessment of AEs were performed by questioning the subject at each scheduled study visit. Treatment Emergent adverse events were defined as any AE during the study that began on or after the date of first dose of investigational product (i.e., Prolastin-C).
Arm/Group | 60 mg/kg Prolastin-C | 120 mg/kg Prolastin-C
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 15/30 | 10/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 60 mg/kg Prolastin-C (N=30) | 120 mg/kg Prolastin-C (N=30)
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 5 (6) — This study used the American Thoracic Society (ATS)/European Respiratory Society (ERS) Task Force definition of exacerbation.
Urinary Tract Infection (Infections and infestations) | 3 (4) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Proteinuria (Renal and urinary disorders) | 2 (2) | 1 (1)
Blood Creatinine Increased (Investigations) | 0 (0) | 2 (2)
Blood Glucose Increased (Investigations) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other